CLINICAL TRIAL: NCT05475613
Title: A Prospective, Single-arm Study of Downstaging Protocol Containing Immunotherapy for HCC Beyond the Milan Criteria Before Liver Transplantation
Brief Title: Downstaging Protocol Containing Immunotherapy for HCC Beyond the Milan Criteria Before Liver Transplantation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2022-145-01
Record Dates: First submitted 2022-07-24; First posted 2022-07-27 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Liver Transplantation; Hepatocellular Carcinoma
Keywords: Liver transplantation; Hepatocellular Carcinoma; Milan Criteria; Downstaging therapy; Locoregional therapies; Targeted therapy; PD1 inhibitor
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Liver Transplantation

STUDY DESIGN:
Intervention Model Description: Eligible patients will undergo downstaging treatment containing an Anti-PD-1 inhibitor (tislelizumab, pembrolizumab, nivolumab et al.). The anti-PD-1 inhibitor will be given intravenously every 3-4 weeks. Other combination regimens, such as locoregional therapies and targeted therapies, will be given to patients according to the protocol decided by the multidisciplinary team of Centers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Downstaging group (Experimental): Eligible patients (See inclusion and exclusion criteria) will undergo downstaging treatment containing Anti-PD-1 inhibitor (tislelizumab, pembrolizumab, nivolumab et al). Anti-PD-1 inhibitor will be given every 3-4 weeks intravenously. Other combination regimens, such as locoregional therapies and targeted therapies will be given to patients according to the protocol decided by the multidisciplinary team of Centers. Patients that have reached the Criteria for Successful Downstage within 12 cycles of downstaging treatment will proceed to the observation phase, while those who fail to meet the Criteria for Successful Downstage after the maximum length of downstaging procedures will drop out from the study.
  Interventions: Procedure: Downstaging procedures containing immunotherapy; Procedure: Liver transplantation

INTERVENTIONS:
Procedure: Downstaging procedures containing immunotherapy — Anti-PD-1 inhibitor will be given every 3-4 weeks intravenously according to the manufacturer's instruction. Other combination regimens, such as locoregional therapies or targeted therapies will be given to patients according to the protocol decided by the multidisciplinary team of Centers.
Procedure: Liver transplantation — Patients with successful downstaging therapy at the end of the observation phase will enroll and undergo liver transplantation unless major medical or oncological contraindications should occur during the waiting phase.

SUMMARY:
Hepatocellular Carcinoma (HCC) is the most common liver malignancy and the third leading cause of cancer death worldwide. Due to the shortage of donor organs and the risk of tumor recurrence after transplantation, the restrictive Milan criteria is the standard guideline for liver transplantation (LT) in patients with HCC and liver cirrhosis. The XXL study (Mazzaferro et al, 2020) is the first prospective trial validating that effective and sustained downstage therapy could expand the selection criteria and improve the prognosis of recipients with HCC beyond Milan criteria. However, the optimal DT protocol is poorly defined, especially in the Asian population. Recently, immunotherapies such as immune-checkpoint inhibitors (ICIs) are revolutionizing the management of advanced HCC, the combination of the ICI and other treatment regimens (Anti-VEGF, locoregional therapies et al) produced superior results in patients with advanced-stage HCC compared to those with traditional therapeutic regimens. Therefore, we hypothesize an intensive downstage regimen containing immunotherapy could expand the selection criteria for HCC LT

DETAILED DESCRIPTION:
This will be a single-arm, open-label, non-randomized phase II study aiming to access the efficacy and safety of the downstage protocol containing immunotherapy for HCC beyond Milan Criteria. This study contains 4 phases:

1. Screening and Downstaging phase Eligible patients (See inclusion and exclusion criteria) will undergo downstaging treatment containing Anti-PD-1 inhibitor (tislelizumab, pembrolizumab, nivolumab et al). Anti-PD-1 inhibitor will be given every 3-4 weeks intravenously. Other combination regimens, such as locoregional therapies and targeted therapies will be given to patients according to the protocol decided by the multidisciplinary team of Centers. Patients that have reached the Criteria for Successful Downstage within 12 cycles of downstaging treatment will proceed to the observation phase, while those who fail to meet the Criteria for Successful Downstage after the maximum length of downstaging procedures will drop out from the study.

   Criteria for Successful Downstage

   Patients that meet 1-4 criteria are considered to have achieved the downstaging goal, otherwise, the downstaging treatment is considered to have failed within 12 cycles of downstaging treatment:
   * CR or PR evaluated by iRECIST/mRECIST after at least 2 cycles of downstaging treatment.
   * Patients with onset AFP<400ng/ml: AFP <400ng/ml at the end of downstaging therapy; Patients with onset AFP>400ng/ml: AFP levels decrease more than 30%, and must be less than 1000ng/ml at the end of downstage therapy.
   * Estimated 5-year overall survival ≥60% at the end of downstaging therapy according to the Metroticket model (http://www.hcc-olt-metroticket.org/calculator).
   * For patients with portal vein tumor thrombus (PVTT1-3), tumor thrombus needs to retract above the bifurcation of the main portal vein, and portal vein anastomosis is feasible during liver transplantation according to the surgeons' judgment.
2. Observation phase Patients that have reached the Criteria for Successful Downstage within 12 cycles of downstaging treatment will proceed to the observation phase ≥ 3 months. Patients at this phase can optionally receive TKIs (sorafenib, lenvatinib et al), and other anti-tumor treatments (such as locoregional therapies, surgery, and immunotherapies et al) are not allowed at this phase. Patients with a sustained response and whose tumors still meet the Criteria for Successful Downstage at the end of the observation phase will be enrolled in the waiting list for liver transplantation, while patients with tumor progression (PD) and their tumors fail to meet the Criteria for Successful Downstage at the end of observation phase will drop out from the study.
3. Waiting and Bridging phase During the waiting period before liver transplantation, patients can optionally receive a non-immunotherapy protocol as bridging treatment determined by the multidisciplinary team (MDT). Surgery is not allowed at this phase.
4. Liver transplantation and post-transplantation phase Patients will undergo liver transplantation unless major medical or oncological contraindications should occur during the waiting phase.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained prior to any screening procedures. Willing and able to comply with scheduled visits, treatment plan and laboratory tests.
2. Patients must have pathologically or cytologically or by radiological criteria proven hepatocellular carcinoma based on the AASLD practice guidelines
3. Patients with HCC must be beyond Milan criteria without extrahepatic metastases or lymph node metastases:

   3.1 Patients without previous treatment: Barcelona clinic liver cancer B-C (China liver cancer stage IIb-IIIa) HCC with or without portal vein tumor thrombus (PVTT 1-3 according to Japanese Vp classification).

   3.2 Patients with late recurrent HCC: The recurrent HCC must be identified no less than 2 years after primary curative treatment (Resection or Radiofrequency, et al), and the recurrent lesions must be localized in the liver and beyond Milan criteria.

   3.3 Patients with early recurrent HCC: The recurrent HCC must be identified within 2 years after primary curative treatment (R0 resection or radiofrequency, et al), and the primary tumor must be within Milan criteria, and the accumulating tumor burden(Primary tumor plus recurrent tumor) must be beyond Milan criteria.
4. Child-Pugh score≤7, with no encephalopathy. Ascites that diuretics can control are permitted in this study.
5. Eastern Cooperative Oncology Group (ECOG) Scale for Assessment of Patient Performance Status (PS score) ≤ 2; KPS score ≥60.
6. Have not received any immunotherapies 6 months before enrollment.
7. Adequate bone marrow, liver, and renal function.
8. The estimated survival before liver transplantation must be more than 12 weeks (Based on the Model for end-stage liver disease, MELD).
9. No other lethal malignancy outside the liver in the past 5 years, such as leukemia, lung cancer, melanoma, etc.
10. Patients with a history of hypertension should be well-controlled (< 140/90 mmHg) on a regimen of anti-hypertensive therapy.
11. Both men and women enrolled in this trial must use adequate barrier birth control measures during the trial and 6 months after the completion of the trial.
12. Patients voluntarily joined the study and signed informed consent with good compliance and follow-up.

Exclusion Criteria

Participants who meet any of the following criteria are not eligible for this study:

1. Histologically/cytologically confirmed cholangiocellular carcinoma, mixed-type liver cancer, or other rare types of liver cancer;
2. Recurrent liver cancer with inadequate initial treatment (i.e., no complete remission or R0 resection);
3. Presence of uncontrollable systemic infections, alcoholism or drug abuse, organic diseases of the heart, lungs, or brain, uncontrolled psychiatric disorders, severe mental illnesses, HIV infection, active tuberculosis, etc.;
4. Presence of severe portal hypertension with a high bleeding risk as assessed by the investigator;
5. History of bleeding events due to portal hypertension in the past 6 months;
6. History of any life-threatening event in the past 6 months, including but not limited to acute myocardial infarction, unstable angina, congestive heart failure, cerebrovascular accidents, pulmonary embolism, major bleeding from other sites, etc.;
7. Severe splenomegaly or splenomegaly-induced neutropenia (ANC < 1.5 × 10⁹/L) or thrombocytopenia (platelet count < 50 × 10⁹/L);
8. History of grade III hepatic encephalopathy or clinical symptoms requiring long-term drainage of pleural effusion, ascites, pericardial effusion, etc.;
9. Uncontrolled hypertension, history of hypertensive crisis or hypertensive encephalopathy;
10. Severe pulmonary hypertension that cannot be controlled by medication;
11. Severe coagulopathy, or those receiving thrombolytic treatment or requiring continuous anticoagulant or antiplatelet therapy for any reason;
12. History of autoimmune diseases such as rheumatoid arthritis, lupus, psoriasis, Crohn's disease, ulcerative colitis, etc.;
13. Major surgical procedure within 4 weeks before the first dose; History of severe allergy to any of the study drugs;
14. Female patients who are pregnant or breastfeeding;
15. Presence of severe psychiatric or psychological disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
For patients with liver transplantation: The 2-year event-free survival rate | 2 years
  From the date of transplantation to the date of tumor recurrence or the date of tumor progression otherwise, with censoring at the date of death or last contact for event-free patients.

SECONDARY OUTCOMES:
For patients with liver transplantation: The 2-year overall survival | 2 years
  The time elapsed from the liver transplantation to death during the 2-year follow-up period.
For all patients with HCC downstaging: 1, 2 year overall survival rate | 1, 2 years
  The probability of survival from the beginning of treatment to the end of 1-year and 2-year follow-up.
For patients with liver transplantation: Rate of early allograft dysfunction (EAD) | 1 week posttransplantation
  Number of recipients developing EAD after liver transplantation
For patients with liver transplantation: Rate of allograft rejection | 1 year
  Number of recipients developing allograft rejection after liver transplantation
For all patients with HCC downstaging: Rate of successful tumor downstaging | 1 year
  Number of patients reaching the successful downstaging criteria for liver transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Chao LIU, PhD, Principal Investigator — Department of Biliary and Pancreatic Surgery, Sun Yat-sen Memorial Hospital, Sun Yat-sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mazzaferro V, Citterio D, Bhoori S, Bongini M, Miceli R, De Carlis L, Colledan M, Salizzoni M, Romagnoli R, Antonelli B, Vivarelli M, Tisone G, Rossi M, Gruttadauria S, Di Sandro S, De Carlis R, Luca MG, De Giorgio M, Mirabella S, Belli L, Fagiuoli S, Martini S, Iavarone M, Svegliati Baroni G, Angelico M, Ginanni Corradini S, Volpes R, Mariani L, Regalia E, Flores M, Droz Dit Busset M, Sposito C. Liver transplantation in hepatocellular carcinoma after tumour downstaging (XXL): a randomised, controlled, phase 2b/3 trial. Lancet Oncol. 2020 Jul;21(7):947-956. doi: 10.1016/S1470-2045(20)30224-2. PMID 32615109
- [Background] Schwacha-Eipper B, Minciuna I, Banz V, Dufour JF. Immunotherapy as a Downstaging Therapy for Liver Transplantation. Hepatology. 2020 Oct;72(4):1488-1490. doi: 10.1002/hep.31234. No abstract available. PMID 32171041
- [Background] Sangro B, Sarobe P, Hervas-Stubbs S, Melero I. Advances in immunotherapy for hepatocellular carcinoma. Nat Rev Gastroenterol Hepatol. 2021 Aug;18(8):525-543. doi: 10.1038/s41575-021-00438-0. Epub 2021 Apr 13. PMID 33850328
- [Background] Tran NH, Munoz S, Thompson S, Hallemeier CL, Bruix J. Hepatocellular carcinoma downstaging for liver transplantation in the era of systemic combined therapy with anti-VEGF/TKI and immunotherapy. Hepatology. 2022 Oct;76(4):1203-1218. doi: 10.1002/hep.32613. Epub 2022 Jul 30. PMID 35765265
- [Background] Tan DJH, Lim WH, Yong JN, Ng CH, Muthiah MD, Tan EX, Xiao J, Lim SY, Pin Tang AS, Pan XH, Kabir T, Bonney GK, Sundar R, Syn N, Kim BK, Dan YY, Noureddin M, Loomba R, Huang DQ. UNOS Down-Staging Criteria for Liver Transplantation of Hepatocellular Carcinoma: Systematic Review and Meta-Analysis of 25 Studies. Clin Gastroenterol Hepatol. 2023 Jun;21(6):1475-1484. doi: 10.1016/j.cgh.2022.02.018. Epub 2022 Feb 16. PMID 35181565
- [Background] Tabrizian P, Holzner ML, Mehta N, Halazun K, Agopian VG, Yao F, Busuttil RW, Roberts J, Emond JC, Samstein B, Brown RS Jr, Najjar M, Chapman WC, Doyle MM, Florman SS, Schwartz ME, Llovet JM. Ten-Year Outcomes of Liver Transplant and Downstaging for Hepatocellular Carcinoma. JAMA Surg. 2022 Sep 1;157(9):779-788. doi: 10.1001/jamasurg.2022.2800. PMID 35857294